CLINICAL TRIAL: NCT05257538
Title: Fecal Microbiota Transplantation in Initial Clostridioides Difficile Enteritis: a Randomized, Placebo-controlled Trial
Brief Title: FMT in Initial CDI
Acronym: FinCDI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Satakunta Central Hospital (Other); Helsinki University Central Hospital (Other); PaijatHame Central Hospital (Other)
Responsible Party: Principal Investigator, Teppo Stenholm, Specialist in gastroenterology and internal medicine, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T123/2021
Record Dates: First submitted 2022-01-27; First posted 2022-02-25 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Clostridioides Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FMT enema (Active Comparator): FMT enema 3-5 days after standard antibiotic treatment
  Interventions: Other: FMT
- plasebo enema (Placebo Comparator): placebo
  Interventions: Other: placebo enema

INTERVENTIONS:
Other: FMT — Fecal microbiota transfer from a healthy and tested volunteer
  Arms: FMT enema
Other: placebo enema — colored water enema
  Arms: plasebo enema

SUMMARY:
The study explores fecal microbiota transfer via retention enema after the first clostridioides difficile episode.

DETAILED DESCRIPTION:
Clostridioides difficile infections (CDI) remain a significant burden for the patients and the society. According to the National Institute for Health and Welfare (THL), in 2018 there were 4324 CDIs in Finland. C. difficile typically affects patients whose gut microbiota is profoundly damaged by antibiotics. Standard therapy for CDI is antibiotic such as vancomycin. After the standard therapy gut microbiota remains damaged and vulnerable to C difficile reinfection arising from spores that survived the treatment. Early recurrence of CDI is commonly defined as relapse of symptoms and positive testing for fecal C difficile within three months after the previous episode. Recurrent CDI is reported in 10-30% of patients after initial treatment, with recurrence approaching 60% after the third episode.

Fecal microbiota transplantation (FMT) is currently the most effective treatment for recurrent CDI (rCDI), with efficacy of over 90%. Even though FMT is mostly administered endoscopically, it is considered a cost-effective way to treat rCDI patients. FMT is recommended after the second relapse, in other words, after the third antibiotic course for CDI. FMT is most effective in rCDI when administered via colonoscopy. However, colonoscopy is a costly and invasive procedure. The largest study exploring a simple and inexpensive retention enema FMT for rCDI showed a 62% clinical response following a single FMT, and 85% after the second. Baro et al. found that FMT via enema was the most cost-effective initial strategy for the management of second recurrence of community-onset CDI.

In the controlled FMT trials the adverse events have been similar with placebo. Also, the long term safety in up to four years follow up seems to be good. The patients treated with FMT seem to normalize their bowel symptoms faster compared to CDI patients treated with only antibiotics.

FMT reduces antibiotic resistance genes in gut microbiota and therefore has a theoretical potential to reduce infections caused by multi-resistant organisms.

A balanced gut microbiota is important in infection control and essential to normal bowel function. CDI is an indicator of damaged gut microbiota. After a course of antibiotics, the gut microbiota typically becomes less diverse for at least some months. It is not known whether the gut microbiota ever regains its former constitution after such a treatment. We hypothesize that planting a new microbial population soon after antibiotic treatment for CDI reduces the risk of recurrence as well as post-infectious functional bowel disorders.

FMT via colonoscopy is currently recommended after the third CDI (second relapse). Our study explores FMT via inexpensive and minimally invasive retention enema after the first CDI episode.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* C. difficile PCR in feces positive and clinical symptoms of enteritis.
* Full resolution of diarrhea during antibiotic treatment for C. difficile
* No other ongoing antibacterial treatments.
* No ongoing probiotics.
* Signed informed consent.

Exclusion Criteria:

* Pregnant
* Ongoing need for antibacterial treatment
* Life expectancy < 1 year
* Prior C. difficile infection in preceding 3 months
* Unable to provide written consent, due to dementia for example.
* Fecal incontinence i.e. inability to retain enema.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
clostridioides difficile relapse rate | month 3

SECONDARY OUTCOMES:
Resolution of gastrointestinal symptoms | month 3 and 1 year
  Primary symptoms of clostridioides difficile infection
composition of fecal microbiota | month 3 and 1 year
  Characterization of fecal microbiome samples down to species level by polymerase chain reaction (PCR)
Retention time, i.e. time from FMT to subsequent defecation | day 1
Fecal microbiota transfer adverse events | within 1 year of administration
  possibly transferred infections, complications of administration etc
Adherence to FMT | From recruitment until FMT administration. Up to 15 days
Alterations in mood as measured by total score of BDI | month 3 and 1 year
  0 to >30 points with higher points meaning more severe depression
Anxiety as measured by total score of GAD-7 | month 3 and 1 year
  0 to 21 points with higher points meaning more severe anxiety
Quality of life as measured by 15D instrument | month 3 and 1 year
clostridioides difficile relapse rate | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No